CLINICAL TRIAL: NCT05950841
Title: A Randomised, Double-blind Study to Determine the Safety and Efficacy of IHAT in Iron Deficient Premenopausal Women.
Brief Title: Safety and Effectiveness of IHAT in Iron Deficient Pre-menopausal Woman
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Nemysis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHATID
Record Dates: First submitted 2023-06-03; First posted 2023-07-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-08

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — locust bean gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose IHAT (Experimental): IHAT in capsule form and carob flour in capsule form - taken as 1 x 100mg IHAT capsule (equiv 30mg iron) in the morning with water and 1 x placebo capsule in the evening with water
  Interventions: Drug: Low dose IHAT
- High dose IHAT (Experimental): IHAT in capsule form - taken as 2 x 100mg (equiv 60mg iron) daily with water (1 in the morning and 1 in the evening)
  Interventions: Drug: High Dose IHAT
- Carob flour (Placebo Comparator): Carob flour in capsule form - taken as 2 x capsules daily with water (1 in the morning and 1 in the evening)
  Interventions: Drug: Carob flour

INTERVENTIONS:
Drug: Low dose IHAT — Once daily dose of 1 capsule (100mg per capsule IHAT) and Once daily dose of 1 capsule (carob flour)
  Arms: Low dose IHAT
Drug: High Dose IHAT — Twice daily dose of 1 capsule (100mg per capsule IHAT)
  Arms: High dose IHAT
Drug: Carob flour — Twice daily dose of 1 capsule (carob flour)
  Arms: Carob flour

SUMMARY:
This is a double blind, randomised, placebo-controlled trial to evaluate orally-dosed IHAT (iron hydroxide adipate tartrate) at 2 different doses compared to placebo for increasing serum ferritin levels in iron-deficient but otherwise healthy premenopausal women over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy iron deficient pre-menopausal women
* Iron deficiency defined as Serum ferritin < 30 ug/L (1)
* Generally healthy defined as C-reactive protein < 3 mg/L (1)
* Subjects adhering to a vegetarian or vegan diet are allowed
* Agree not to give blood donations during the study
* Able to provide informed consent
* Agree not to participate in another clinical trial while enrolled in this trial
* Agree not to change current diet and/or exercise frequency or intensity

Exclusion Criteria:

* Anaemia (as determined from the haematocrit and haemoglobin measures) (2)
* Previously told they have an iron absorption problem
* Subjects regularly taking iron specific supplements during or 2 months prior to study commencement (the use of other mineral/vitamin/herbal preparations is allowed but should be recorded) (3)
* Any uncontrolled serious illness (4)
* Receiving/prescribed coumadin (Warfarin), heparin, dalteparin, enoxaparin or other anticoagulation therapy
* Active smokers, nicotine use, alcohol(5) or drug (prescription or illegal substances) abuse
* Chronic gastrointestinal disorders
* Pregnant/lactating women or women trying to conceive
* Diagnosed depression or mental disorder that is uncontrolled
* Eating disorders
* BMI > 35 kg/m2
* Allergic to any of the ingredients in active or placebo formula
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other clinical trial during the past 1 month

Footnotes

1. A blood test is required prior to enrolment into the study to receive trial product. Participants will be required to attend a local pathology collection centre and have serum ferritin and CRP within the required limits to be considered enrolled in the study and be provided with trial product.
2. Anyone considered to be anaemic will be excluded and directed to their GP. In women, anaemia is defined as any of the following: Haemoglobin < 115 g/L, Haematocrit < 35%.
3. Potential participants that are taking supplements that would result in their exclusion must wait an 8-week washout period prior to commencing the study.
4. An uncontrolled illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
5. Chronic past and/or current alcohol use (>14 alcohol drinks/week).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of women recovering from ID at week 12 | Week 12
  Percentage of women recovering from ID at week 12, defined as serum ferritin levels of 30 -150 ug/L

SECONDARY OUTCOMES:
Time to reach normalisation of ferritin levels | Baseline, week 6 and week 12
  Time to reach normalisation of ferritin levels via blood test results
Iron Status | Baseline, week 6 and week 12
  Iron Status (Serum ferritin, Hb levels, Serum iron levels, TSAT levels, NTBI) via blood test
Incidence and prevalence of gastrointestinal side effects | Baseline, weeks 1 - 5, week 6 and week 12
  - Incidence and prevalence of gastrointestinal side effects via Gastrointestinal questionnaire
Change in fatigue | Baseline, week 6 and week 12
  Change in fatigue via Fatigue Severity Questionnaire
Iron deficiency symptoms | Baseline, week 6 and week 12
  Iron deficiency symptoms via SF-36 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, New Farm, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared